CLINICAL TRIAL: NCT06028516
Title: ctDNA Monitoring Cancer Recurrence and Its Clinical Value in Solid Tumor
Brief Title: MRD Application in Colorectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong First Medical University (Other)
Collaborators: Jinan Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Manfei01
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Surgery; Chemotherapy Effect
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We first collect tumor tissue and adjacent tissue to peform the WES sequencing, then collect blood after postoperative surgery 1, 3. 6, 9, 12, 18, 24 month to detect ctDNA.

DETAILED DESCRIPTION:
ctDNA is obtained from plasma rather than serum, as the latter contains more DNA released from immune cells during clotting. Blood should be drawn into a K2EDTA or cell stabilization tube (e.g., Streck cfDNA collection tube). Plasma isolation should be performed as soon as possible, no later than 24 hours, using K2EDTA (preferably within 4-6 hours) and, if using cell stabilization tubes, within 2-7 days, temporarily stored at 4°C.

Sample disposal procedure: collect whole anticoagulated blood, gently invert to fully anticoagulate, plasma fractionation should be performed as soon as possible, no later than 24 hours, temporarily stored at 4°C using K2EDTA (preferably within 4-6 hours), and stored at -80°C for long term. The collected anticoagulant blood is placed in an ice box containing ice packs and transported vertically to a centrifugable laboratory. Centrifuge at 3000 rpm at 4°C for 15 min, take the upper layer, and aliquot 0.5 mL/tube into 1.5 mL centrifuge tubes. Cryopreserved at -80 °C, 1 mL of whole blood yields approximately 0.5 mL of plasma.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with colorectal tumors, whose clinical symptoms meet the diagnostic criteria of colon cancer in my country, and pathologically diagnosed as colorectal cancer after surgery; (2) patients with stage II-III colorectal cancer; (3) aged 30-80 years; (4) All underwent conventional radiotherapy and chemotherapy after operation; (5) Complete clinical data and follow-up records were available.

Exclusion Criteria:

* (1) Other serious diseases (cardiovascular and cerebrovascular diseases, kidney diseases, etc.) before operation; (2) Combined with multiple primary colorectal cancers; (3) Patients with other malignant tumors within the past 5 years; (4) Combined with digestive tract Obstruction, perforation, bleeding and other indications for emergency surgery.

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer and they were received routine laparoscopic surgery and regular chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA positive patients are detedcted before PET-CT | 2023.12.31
  multiple PCR based on the WES results

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xu, PhD, Study Director — Shandong First Medical University
Locations (1):
- Jinan central hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
It will be available when our paper is accepted.

REFERENCES:
- [Background] Zhou J, Wang C, Lin G, Xiao Y, Jia W, Xiao G, Liu Q, Wu B, Wu A, Qiu H, Zhang F, Hu K, Xue H, Shen Z, Wang Z, Han J, Niu B, Xu Y, Yu Z, Yang L. Serial Circulating Tumor DNA in Predicting and Monitoring the Effect of Neoadjuvant Chemoradiotherapy in Patients with Rectal Cancer: A Prospective Multicenter Study. Clin Cancer Res. 2021 Jan 1;27(1):301-310. doi: 10.1158/1078-0432.CCR-20-2299. Epub 2020 Oct 12. PMID 33046514
- [Result] Chen G, Peng J, Xiao Q, Wu HX, Wu X, Wang F, Li L, Ding P, Zhao Q, Li Y, Wang D, Shao Y, Bao H, Pan Z, Ding KF, Cai S, Wang F, Xu RH. Postoperative circulating tumor DNA as markers of recurrence risk in stages II to III colorectal cancer. J Hematol Oncol. 2021 May 17;14(1):80. doi: 10.1186/s13045-021-01089-z. PMID 34001194